CLINICAL TRIAL: NCT04915703
Title: Flushing of Internalized Percutaneous Transhepatic Biliary Drainage Catheters
Acronym: FLUSH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Adriaan Moelker, Radiologist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL77857.078.21
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Bile Duct Obstruction
Keywords: bile duct; obstruction
MeSH Terms: conditions — Cholestasis; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Non-blinded randomized controlled trial with 1:1 allocation
Masking Description: open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): flushing of internal external PTBD catheter 3 times a day
  Interventions: Procedure: Flushing of PTBD catheter
- Standard of Care (No Intervention): no flushing of PTBD catheter

INTERVENTIONS:
Procedure: Flushing of PTBD catheter — flushing of internal external PTBD catheter 3 times a day
  Arms: Intervention

SUMMARY:
Percutaneous transhepatic biliary drainage (PTBD) is a drainage method for biliary obstruction. Patients with a PTBD catheter often need multiple re-interventions because of symptoms of catheter obstruction such as pain, jaundice, pruritus, leakage and/or fever. The onset of these symptoms results in hospital visits, opening of the external catheter of an internal external PTBD and re-interventions.

The investigators hypothesize that daily flushing of an internal external biliary catheter will increase the time-to-symptom-onset.

DETAILED DESCRIPTION:
Bile is synthesized and secreted by the liver and transported into the peripheral bile ducts, to the left or right hepatic duct which join together in the common hepatic duct and more distally in the common bile duct. Secreted bile is stored in the gall bladder. During a meal, the bile is secreted into the duodenum.

Obstruction of the biliary tract will result in cholestasis with symptoms as jaundice and pruritus and cholangitis in case of infection, usually related to prior biliary intervention. Causes of biliary obstruction are benign or malignant.

Percutaneous transhepatic biliary drainage (PTBD) is a drainage method for biliary obstruction. The procedure starts with percutaneous puncture under fluoroscopic or ultrasound guidance and cannulation of the peripheral biliary tree, which is confirmed by contrast injection in the biliary tree. The needle will be exchanged for a guidewire which can be advanced into the biliary tract. When the correct position is reached, a drainage catheter with side holes is placed.

There are two types of PTBD techniques: placement of an external biliary drain and placement of an internal external biliary drain. The external biliary drain is positioned in the bile duct above a stenosis and drains the bile externally into a bag outside the patient. Capping of an external biliary drain will stop the drainage of bile into the bag and forces the bile to drain towards the digestive tract. The internal external biliary drain is placed in the bile duct and the tip of the internal external biliary drain is localised in the duodenum allowing both bile flow through the drain to the digestive tract (internal) or into the bag (external). Capping of an internal external biliary drain will stop the external drainage and results in internal drainage only.

Complications of PTBD are bleeding (usually during or shortly after the procedure), infection (cholangitis, abscess, peritonitis, cholecystitis, pancreatitis), catheter obstruction and catheter dislocation(1). Catheter obstruction will result in cholestasis resulting in jaundice, drain leakage and finally cholangitis. The exact prevalence of PTBD catheter obstruction is not described in literature, however the prevalence of cholangitis in patients with a PTBD catheter is reported as high as 59%(2). Subsequently, the PTBD catheter often needs a revision (re-intervention), i.e. exchanging the catheter for a new one. If catheter obstruction is assessed during re-intervention, attempts can be made to remove the obstruction or the obstructed PTBD catheter can be exchanged for a new PTBD catheter.

After PTBD catheter placement, flushing of the PTBD catheter is not standard protocol in our center. In clinical practice, when obstruction of PTBD catheter occurs, the study team will advise patients to start with daily flushing of the PTBD catheter which the investigators believe will decrease the extent of obstruction and omits re-intervention. The investigators performed a literature search and the investigators did not find any clinical trial on the efficacy of flushing of PTBD catheters. Guidelines of the Society of Interventional Radiology on percutaneous biliary drainage do not mention flushing of the catheter(1). The investigators did find some publications in which an advice with regard to flushing of a PTBD catheter was mentioned, however without any scientific substantiation(3-7).

There is no scientific evidence for or against PTBD catheter flushing. Flushing is a simple, low-cost and low-risk procedure. Complications or side-effects of PTBD catheter flushing are not reported in literature. PTBD re-interventions on the other hand are associated with risks and are invalidating for the patient. The investigators hypothesize that daily flushing of an internal external biliary catheter will increase the time-to-symptom-onset requiring hospital visits and re-interventions in this patient group.

ELIGIBILITY:
Inclusion Criteria:

Patient with obstruction of the bile duct(s) planned for internal external PTBD;

* Proficient in Dutch language;
* Written informed consent.

Exclusion Criteria:

* Age < 18 years;

  * No informed consent;
  * Pregnancy;
  * Obstruction caused by gall stones;
  * External PTBD catheter (without internalization);
  * Patient has already a PTBD catheter;
  * More than 1 PTBD catheter is placed at intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
time-to-symptom-onset in patients with an internal external PTBD catheter without daily flushing compared to patients with an internal external PTBD catheter who daily flush the catheter | 12 weeks
  time-to-symptom-onset

CONTACTS AND LOCATIONS:
Overall Officials: laurens Groenendijk, Study Director — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No